CLINICAL TRIAL: NCT07074769
Title: In-Lab Evaluation of A Hearing Aid Housed in Ophthalmic Spectacles for Mild to Moderate Hearing Loss
Brief Title: Evaluation of In-lab Benefit for Speech-in-noise Intelligibility With Device for Adults With Mild to Moderate Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxottica Group S.p.A. (Industry)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol version 4 9.6.2025
Record Dates: First submitted 2025-06-30; First posted 2025-07-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A prospective in-lab within-subjects design with repeated measures (Experimental): Test of speech recognition in noise (the Matrix test). Assessment of speech recognition in babble (The Connected Speech Test). Device users' ratings of listening effort in noise with and without the device.
  Interventions: Device: Evaluation of speech-in-noise intelligibility and listening effort

INTERVENTIONS:
Device: Evaluation of speech-in-noise intelligibility and listening effort — The speech in noise testing will be performed in lab settings; the listening effort evaluated trough a standardized questionnaire

SUMMARY:
Evaluation of in-lab benefit for speech-in-noise intelligibility with the device for adults with mild to moderate hearing loss.

DETAILED DESCRIPTION:
This primary objective is to evaluate whether the device improves speech recognition in noise compared to the clinically relevant comparison condition of no treatment (unaided) for adults with mild to moderate hearing loss. The primary outcome will be measured using a clinically available test of speech recognition in noise that uses adaptive bracketing of signal to noise ratio (the Matrix test). The secondary outcome will also assess speech recognition in babble at ecologically valid fixed signal to babble ratios (The Connected Speech Test). Tertiary outcomes will examine device users' ratings of listening effort in noise with and without the device.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* symmetrical bilateral mild to moderate sensorineural hearing loss
* native speakers of English.

Exclusion Criteria:

* Children
* those without hearing loss
* those without symmetrical bilateral mild to moderate sensorineural hearing loss
* those who do not wish to wear the test device instead of their own spectacles during the in-lab procedure
* those who are not native speakers of English
* those who have pacemakers, other implantable devices, or insulin pumps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Unaided and Aided speech in noise Matrix test | 1 hour
  Matrix Test with and without device. The outcome is Speech Reception Threshold (SRT) in dB SNR
Unaided and Aided Connected speech-in-noise tests | 1 hour
  Connected Speech Test with and without device. The outcome is the percentage score representing the number of key words correctly repeated

SECONDARY OUTCOMES:
Unaided vs Aided Ratings of Listening Effort | 30 minutes
  Evaluation of the listening effort with and without device trough questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No